CLINICAL TRIAL: NCT01148849
Title: A Phase 1, Dose Escalation Study of MGAH22 in Patients With Refractory HER2 Positive Breast Cancer and Patients With Other HER2 Positive Carcinomas for Whom No Standard Therapy Is Available
Brief Title: Safety Study of MGAH22 in HER2-positive Carcinomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MacroGenics (Industry)
Collaborators: Green Cross Corporation (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-MGAH22-01; 02598-10 (Other Grant/Funding Number: NCI CRADA); NCT01195935 (obsolete NCT alias)
Record Dates: First submitted 2010-06-17; First posted 2010-06-22 (Estimated); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer; Gastric Cancer
MeSH Terms: conditions — Breast Neoplasms; Stomach Neoplasms | interventions — margetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- Cohort 1: 0.1 mg/kg weekly for 4 weeks (Experimental): Anti-HER2 monoclonal antibody (margetuximab)
  Interventions: Biological: margetuximab
- Cohort 2: 0.3 mg/kg weekly for 4 weeks (Experimental): Anti-HER2 monoclonal antibody (margetuximab)
  Interventions: Biological: margetuximab
- Cohort 3: 1.0 mg/kg weekly for 4 weeks (Experimental): Anti-HER2 monoclonal antibody (margetuximab)
  Interventions: Biological: margetuximab
- Cohort 4: 3.0 mg/kg weekly for 4 weeks (Experimental): Anti-HER2 monoclonal antibody (margetuximab)
  Interventions: Biological: margetuximab
- Cohort 5: 6.0 mg/kg weekly for 4 weeks (Experimental): Anti-HER2 monoclonal antibody (margetuximab)
  Interventions: Biological: margetuximab
- Cohort 6: 10 mg/kg weekly every 3 weeks (Experimental): Anti-HER2 monoclonal antibody (margetuximab)
  Interventions: Biological: margetuximab
- Cohort 7: 15 mg/kg weekly every 3 weeks (Experimental): Anti-HER2 monoclonal antibody (margetuximab)
  Interventions: Biological: margetuximab
- Cohort 8: 18 mg/kg weekly every 3 weeks (Experimental): Anti-HER2 monoclonal antibody (margetuximab)
  Interventions: Biological: margetuximab

INTERVENTIONS:
Biological: margetuximab — margetuximab
  Other Names: MGAH22

SUMMARY:
The purpose of this study is to determine if MGAH22 is safe when given by intravenous (IV) infusion to patients with HER2-positive cancer. The study will also evaluate how long MGAH22 stays in the blood and how long it takes for it to leave the body, what is the highest dose that can safely be given, and whether it has an effect on tumors.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed carcinoma that overexpresses HER2 by immunohistochemistry (2+ or 3+ positivity by HercepTest or equivalent).
* Progressive disease during or after last treatment regimen.
* Appropriate treatment history for histological entity.
* ECOG Performance Status <= 1.
* Life expectancy >= 3 month.
* Measurable disease
* Acceptable laboratory parameters and adequate organ reserve.
* Baseline LVEF >50%

Exclusion Criteria:

* Lifetime anthracycline exposure > 350 mg/m2 of doxorubicin or equivalent
* Major surgery within four weeks before enrollment.
* Known hypersensitivity to murine or recombinant proteins, polysorbate 80, or any excipient contained in the drug formulation.
* Second primary malignancy that has not been in remission for greater than 3 years. Treated non-melanoma skin cancer, cervical carcinoma in situ on biopsy, or squamous intraepithelial lesion on PAP smear, localized prostate cancer (Gleason score < 6), or resected melanoma in situ are exceptions and do not require a 3 year remission.
* Active viral, bacterial, or systemic fungal infection requiring parenteral treatment within four weeks of enrollment. Patients requiring any oral antiviral, fungal, or bacterial therapy must have completed treatment within one week of enrollment.
* History of chronic or recurrent infections that require continual use of antiviral, antifungal, or antibacterial agents.
* History of deep vein thrombosis, pulmonary embolism, myocardial infarction, or stroke within three months of enrollment.
* Known history of central nervous system (CNS) metastatic disease with evidence of residual or recurrent disease upon entry.
* New York Heart Association class III or IV heart disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2010-07; Primary Completion 2022-06-14 (Actual); Study Completion 2022-06-14 (Actual)

PRIMARY OUTCOMES:
Occurrence of Adverse Events and Serious Adverse Events | Up to 28 days after last infusion
  Note that serious adverse events that are considered study drug related can be reported at any time after Study Day 50 or 28 days after the last infusion.

SECONDARY OUTCOMES:
Number of participants with dose limiting toxicities for weekly dosing | up to Study Day 28 for weekly dosing
  Characterize maximum tolerated dose (MTD) or maximum administered dose (MAD) (if no MTD is defined) of margetuximab
Number of participants with dose limiting toxicities every 3-week dosing | Up to Study Day 21 day for every 3-week dosing
  Characterize maximum tolerated dose (MTD) or maximum administered dose (MAD) (if no MTD is defined) of margetuximab
Concentration of Margetuximab at Steady State once-weekly doses of margetuximab | Study Day 1, 2, 4, 5, 8, 15, 22, 29 ,36, 50, every 4 weeks thereafter throughout study completion, average 2 months.
Number of patients who develop treatment-emergent anti-drug antibodies to margetuximab (Immunogenicity) | Study Day 1, 22, 50, every 4 weeks thereafter throughout study completion, average 2 months.
Maximum Concentration of Margetuximab at Steady State once every 3 weeks schedule | Study Day 1, 2, 4, 5, 22, 29 ,36, 50, every 3 weeks thereafter throughout study completion, average 10 months.
Area Under the Concentration Time Curve at Steady State (AUC ss) once every 3 weeks schedule | Study Day 1 through Day 22
  AUC is a mathematical calculation that describes the drug concentration in the blood over time.
Area Under the Concentration Time Curve at Steady State (AUC ss) weekly dosing schedule | Study Day 1 through Day 8
  AUC is a mathematical calculation that describes the drug concentration in the blood over time.
Clearance once every 3 weeks schedule | Study Day 1, 2, 4, 5, 22, 29 ,36, 50, every 3 weeks thereafter through study completion, average 10 months
  Drug clearance is the amount of drug removed from the bloodstream per unit of time.
Volume of Distribution at Steady State once every 3 weeks | Study Day 1, 2, 4, 5, 22, 29 ,36, 50, every 3 weeks thereafter through study completion, average 10 months
  The volume of distribution is related to a whether how much drug is distributed to body tissues or remains in the bloodstream
Terminal Half-life once every 3 weeks schedule | Study Day 1 through Day 22
  Terminal half-life is the time required to divide the plasma concentration by two after reaching pseudo-equilibrium.
Terminal Half-life once every weekly dosing schedule | Study Day 1 through Day 8
  Terminal half-life is the time required to divide the plasma concentration by two after reaching pseudo-equilibrium.
Number of Patients Who Develop Treatment-emergent Anti-drug Antibodies to Margetuximab once every 3 weeks schedule | Study Day 1, 2, 4, 5, 22, 29 ,36, 50, every 3 weeks thereafter through study completion, average 10 months
Number of Patients with a Complete Response (CR) or Partial Response (PR) to Treatment | Assessed at 6, 18, 30, 42, and 54 weeks, they every 24 weeks until treatment discontinuation, average 10 months
  Investigate the preliminary anti-tumor activity as measured by response to treatment of margetuximab, using conventional Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
Duration of response | Assessed at 6, 18, 30, 42, and 54 weeks, they every 24 weeks until treatment discontinuation,average 10 months
  Duration of response is calculated at the time from CR or PR to relapse or cancer progression
Progression free survival | Assessed at 6, 18, 30, 42, and 54 weeks, they every 24 weeks until treatment discontinuation, average 10 months
  The interval between the first dose of study medication and progression of disease or death from any cause
Number of patients with complete response, partial response, stable disease, or progressive disease according to each CD16A-158 genotype (FF, FV, VV) | Fc receptor genotypes assessed prior to study treatment. Response to treatment assessed at 6, 18, 30, 42, and 54 weeks, then every 24 weeks until treatment discontinuation, average 10 months
  Fc Receptor polymorphisms may affect responsiveness to immunotherapies
Changes in immune cell subsets | Before infusion and 1 hour after infusion on Study Day 1, Study Day 2, before infusion on Study Day 22 and 50
  Changes in immune cell subsets may affect responsiveness to immunotherapies
Serum cytokines in the blood | Study Day 1, 2, 4, 5, 22, 29 ,36, 50, every 3 weeks thereafter through study completion, average 10 months
  Changes in the levels of cytokines in the blood may be related to an immune response to treatment.
Amount HER2 in the blood | Before infusion and 1 hour after infusion on Study Day 1, Study Day 2, before infusion on Study Day 22 and 50
  Levels of HER2 in the bloodstream may indicate response to treatment.
Antibody dependent cellular cytotoxicity (ADCC) activity | Before infusion and 1 hour after infusion on Study Day 1, Study Day 2, before infusion on Study Day 22 and 50
  ADCC activity is the ability of immune cells (like lymphocytes) to kill cells that have immune markers (like HER2) on the cell surface
Fc receptor occupancy | Before infusion and 1 hour after infusion on Study Day 1, Study Day 2, before infusion on Study Day 22 and 50
  Fc receptor occupancy is the amount of time that the receptor is bound to an immune marker (like HER2) on the cell surface.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - National Cancer Institute, Bethesda, Maryland
  - Sarah Cannon Research Institute, Nashville, Tennessee
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Bang YJ, Giaccone G, Im SA, Oh DY, Bauer TM, Nordstrom JL, Li H, Chichili GR, Moore PA, Hong S, Stewart SJ, Baughman JE, Lechleider RJ, Burris HA. First-in-human phase 1 study of margetuximab (MGAH22), an Fc-modified chimeric monoclonal antibody, in patients with HER2-positive advanced solid tumors. Ann Oncol. 2017 Apr 1;28(4):855-861. doi: 10.1093/annonc/mdx002. PMID 28119295